CLINICAL TRIAL: NCT01660074
Title: Glycemic Index and Glycemic Response of Food and Products That Produced in Taiwan
Brief Title: Glycemic Index and Glycemic Response of Food and Products
Acronym: GI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Pingtung University Science and Technology (Other)
Responsible Party: Principal Investigator, Lin Meng Hsueh Amanda Lin, PostDoc, National Pingtung University Science and Technology
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: FP202
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: glycemic index, resistant starch, glycemic response
MeSH Terms: interventions — Resistant Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test food, reference food (Experimental): Test food group of subject need to comsume 50g available carbohydrate of test food. One test food for one ocassion. Reference food need to comsume same 50g available carbohydrate of reference food, usually white bread or glucose syrup.
  Interventions: Other: test food

INTERVENTIONS:
Other: test food — All food, include reference food was tested in 50g available carbohydrate portion size.
  Other Names: Starchy food; Taiwan local fruits; White bread; White bread with resistant starch

SUMMARY:
The purpose of ths study was to evaluate the glycemic index and glycemic response of food and products that produced in Tiwan. The food and product are in includes local produced fruits, starchy food and bread made from resistant starch.

DETAILED DESCRIPTION:
Low glycemic index (GI) diets have protective and therapeutic potential for diabetic patients and general public. With recent recognition of resistant starch (RS), an indigestible fraction which has postprandial glucose lowering effects, the addition of resistant starch in bread may alter its glycemic effects and thus glycemic index. Therefore, the objectives of this study were to investigate the glycemic index, glycemic reponse of Taiwan local food and effects of resistant starch in bread formulation.

ELIGIBILITY:
Inclusion Criteria:

* 1) healthy weight, stable for 6 months prior to the study, 2) not being on a diet, 3) not taking prescription medication, 4) not a smoker, 5) normotensive and 6) normal fasting glucose

Exclusion Criteria:

-

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
glycemic index | 2 hour postprandial blood glucose
  White bread was the reference food (GI = 100%) against which all test foods were compared. Subjects arrived at the laboratory at eight to nine o'clock in the morning after 10-12 h overnight fast. Each subject was fed equivalent 50 g available carbohydrate of test foods or reference food in random order. To minimize day to day variation of glucose tolerance, the reference food was tested in triplicate in each subject. All test and reference foods were served with 220 mL of water. An automatic lancet device (Safe-T-Pro Diagnostics GmbH Mannheim, Germany) was used to collect finger capillary blood samples (1.5 mL). Blood samples were taken immediately before the start of the study (0 min) and 15, 30, 45, 60, 90 and 120 min after the start of eating.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Meng-Hsueh, PhD, Principal Investigator — NPUST
Locations (1):
- Food Science Department, Pingtung City, Taiwan

REFERENCES:
- See also: Glycemic index research institute — http://www.glycemic.com/
- See also: GI research University of Sydney — http://www.glycemicindex.com/